CLINICAL TRIAL: NCT05324423
Title: A Single-center, Open-access Study to Evaluate Drug Interactions Between XNW3009, Febuxostat, and Colchicine in Patients With Gout
Brief Title: To Evaluate Drug Interactions Between XNW3009, Febuxostat, and Colchicine in Patients With Gout
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW3009-I-04
Record Dates: First submitted 2021-12-12; First posted 2022-04-12 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Other): Colchicine 0.5 mg Oral Tablet Day-7~Day25 qd, Febuxostat 40 mg Oral Tablet Day1 and Day14 qd, XNW3009 0.5 mg Oral Tablet Day8~Day21 qd.
  Interventions:
  Drug: Colchicine Drug: Febuxostat Drug: XNW3009
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine0.5 mg Oral Tablet Day-7~Day25 qd；Febuxostat 40 mg Oral Tablet Day1 and Day14 qd；XNW3009 0.5 mg Oral Tablet Day8 and Day21 qd
  Other Names: Febuxostat、XNW3009

SUMMARY:
A single-center, open-access study to evaluate drug interactions between XNW3009, febuxostat, and colchicine in patients with gout

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥18.0 and ≤32 kg/m2;
* Screening sUA value ≥480μmol/L;
* Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination，imaging examination or safety laboratory values.

Exclusion Criteria:

* Subject known or suspected of being sensitive to the study drugs or its ingredient；sCr>ULN；
* History of kidney stones or screening kidney stones by B-ultrasound;
* History of malignancy；
* History of xanthinuria；
* Donated blood（≥400ml）within 3 months prior to screening or received transfusion of blood
* ALT or AST > 1.5 x ULN
* Unstable angina, history of symptomatic arrhythmia, or heart failure
* HbAlc>8%
* eGFR<60ml/min/1.73m2
* Investigational drug within 3 months of study dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Observed maximum concentration at steady state (Cmax,ss) | 100 days
  To evaluate the maximum concentration at steady state of oral XNW3009 tablets, febuxostat, and colchicine in patients with gout
Observed area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) | 100 days
  To evaluate the AUCss of oral XNW3009 tablets, febuxostat, and colchicine in patients with gout

SECONDARY OUTCOMES:
Time to Maximum Serum Concentration (Tmax) | 100 days
  To evaluate the Tmax of oral XNW3009 tablets, febuxostat and colchicine in patients with gout
Mean Terminal Phase Half-life (t1/2) | 100 days
  To evaluate the t1/2 of XNW3009 tablets, febuxostat and colchicine in gout patients
Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) | 100 days
  Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Serum or urine Uric Acid Level | 100 days
  Change in Serum or urine Uric Acid Level
Serum or urine Creatinine | 100 days
  Change in Serum or urine Creatinine
Number of Participants With Clinically Significant Laboratory Test Abnormalities | 100 days
  Investigator judged clinical significance of laboratory test abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Xu, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No